CLINICAL TRIAL: NCT04554485
Title: Single Cycle of Blinatumomab Followed by High-dose Chemotherapy in the Induction Therapy for Ph-negative Acute Lymphoblastic Leukemia in Adults
Brief Title: Blinatumomab Followed by High-dose Chemotherapy for Ph-negative Acute Lymphoblastic Leukemia (ALL)
Acronym: Blina-CELL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology and Blood Transfusion, Czech Republic (Other)
Collaborators: CZECRIN - Czech Clinical Research Infrastructure Network (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Blina-CELL
Record Dates: First submitted 2020-09-07; First posted 2020-09-18 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2023-09

CONDITIONS: Lymphoblastic Leukemia, Acute, Adult; Ph Negative ALL; Newly Diagnosed
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blinatumomab followed by high-dose chemotherapy (Experimental): Single cycle of blinatumomab followed by high-dose chemotherapy in the induction therapy for Ph-negative acute lymphoblastic leukemia in adults
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Single cycle of blinatumomab followed by high-dose chemotherapy in the induction therapy for Ph-negative acute lymphoblastic leukemia in adults
  Other Names: BLINCYTO; AMG103; L01XC19

SUMMARY:
This is a phase II interventional trial to evaluate the efficacy of blinatumomab followed by high-dose chemotherapy in the first-line treatment for Ph-negative acute lymphoblastic leukemia (ALL) in adults. The aim is to increase the number of complete molecular responses after first two cycles of therapy. Early molecular response is considered to be the most powerful prognostic factor in ALL. Thus, a higher proportion of early molecular responses should translate into improved survival and fewer indications for allogeneic stem cell transplants

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the percentage of complete molecular responses after two cycles of induction therapy composed of a single cycle of blinatumomab followed by chemotherapy. Molecular response id monitored by a patient-specific Ig/TCR rearrangements in an assay with the sensitivity of at least 10e-04.

Outline:

Run-in phase: dexamethasone 10 mg/m2 PO (day 1-7), cyclophosphamide IV 200 mg/m2 (day 3-5), vincristine 2 mg IV (day 6), daunorubicin 45 mg/m2 IV (day 6-7), G-CSF until recovery, methotrexate 15 mg IT.

Day 11: Screening to the study. Induction I: blinatumomab 9 µg/day IV continuously (day 12-19), dose step to 28 µg/day (day 19-40). Induction II: dexamethasone 10 mg/m2 PO (day 50-54), vindesine 3 mg/m2 IV (day 50), methotrexate 1.5 g/m2 IV (day 50), etoposide 250 mg/m2 IV (day 53-54), cytarabine 2x 2 g/m2 IV (day 54), G-CSF until recovery, methotrexate 15 mg + cytarabine 40 mg + dexamethasone 4 mg IT (day 60).

Week 11: Primary endpoint assessment.

* Complete Remission (CR) and Complete Remission with incomplete blood count recovery(CRi) continue with Consolidation I;
* no CR/CRi: end of study, salvage regimen upon the investigator´s decision.

Consolidation I (week 13): rituximab 375 mg/ m2 IV (day 0, if CD20+ at diagnosis), methotrexate 1.5 g/m2 IV (day 1, 15), PEG-asparaginase 2000 U/m2 IV (day 2, 16), 6-MP 60 mg/m2 PO (day 1-7, 15-21), methotrexate 15 mg + cytarabine 40 mg + dexamethasone 4 mg IT (day 1).

Week 18 assessment:

* CR/CRi and MRD <10-4: continue the protocol;
* CR/CRi and MRD ≥10-4;

  * and CR/CRi on day 40 or ≥50% reduction of bone marrow blasts on day 40: 1-2 cycles of blinatumomab followed by alloSCT;
  * and no CR/CRi on day 40 and <50% reduction of bone marrow blasts on day 40: 1 cycle of high dose chemotherapy followed by alloSCT;
* relapse: end of study.

Consolidation II (week 19): rituximab 375 mg/ m2 IV (day 0, if CD20+ at diagnosis), prednisone 60 mg/m2 PO (day 1-14), vindesine 3 mg/m2 IV (day 1, 7), adriamycine 50 mg/m2 IV (day 1, 7), cyclophosphamide 1000 mg/m2 IV (day 15), cytarabine 75 mg/m2 IV (day 17-20, 24-27), thioguanine 60 mg/m2 PO (day 15-28), methotrexate 15 mg + cytarabine 40 mg + dexamethasone 4 mg IT (day 1), methotrexate 15 mg IT (day 17, 24). Consolidation III+VI (week 27 and 43): rituximab 375 mg/ m2 IV (day 0, if CD20+ at diagnosis), methotrexate 1.5 g/m2 IV (day 1, 15), PEG-asparaginase 2000 U/m2 IV (day 2, 16), 6-MP 60 mg/m2 PO (day 1-7, 15-21). Consolidation IV (week 33): rituximab 375 mg/ m2 IV (day 0, if CD20+ at diagnosis), cytarabine 1000 mg/m2 IV (day 1, 3, 5), methotrexate 15 mg + cytarabine 40 mg + dexamethasone 4 mg IT (day 8). Consolidation V (week 38): rituximab 375 mg/ m2 IV (day 0, if CD20+ at diagnosis), cyclophosphamide 1000 mg/m2 IV (day 1), cytarabine 500 mg/m2 IV (day 1), methotrexate 15 mg + cytarabine 40 mg + dexamethasone 4 mg IT (day 1).

Maintenance (start at week 49, duration 12 months): 6-MP 60 mg/m2 PO daily, methotrexate 20 mg/m2 weekly.

(Doses of daunorubicin, methotrexate, cytarabine and PEG-asparaginase are reduced in patients >55 years.)

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years;
* Lymphoblasts positive for CD19;
* Eligible to intensive chemotherapy, due to general health status;
* With newly diagnosed B-precursor-ALL;
* Without BCR-ABL fusion by FISH analysis and/or RT-PCR;
* Blasts expressing the CD19 antigen by flow cytometry;
* Previously untreated;
* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2;
* Diagnostic sample of bone marrow (or peripheral blood with >50% of blasts) available for central MRD assessment
* Written informed consent obtained prior to any screening procedures.

Exclusion Criteria:

* History of malignancy other than ALL within 5 years prior to start of protocol-required therapy, except for:

  * Malignancy treated with curative intent and with no known active disease present for 5 years before enrollment and felt to be at low risk for recurrence by the treating physician;
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease;
  * Adequately treated cervical carcinoma in situ without evidence of disease;
  * Adequately treated breast ductal carcinoma in situ without evidence of disease;
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer.
* History or presence of central nervous system (CNS) pathology as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis;
* Persisting ALL in the CNS at the end of run-in period; patients with initial cerebrospinal fluid (CSF) infiltration arriving into CSF negativity after up to 4 intrathecal applications of chemotherapy within the first 10 days of therapy are allowed for the study;
* Current autoimmune disease or history of autoimmune disease with potential CNS involvement;
* Active known hepatitis B virus (HBV) or hepatitis C virus (HCV) or positive HIV serology;
* Hypersensitivity to any active substance contained in blinatumomab, including polysorbate 80;
* Vaccination with a live virus vaccine within 4 weeks prior to the study enrolment;
* Female patients who are pregnant or breast feeding or patients of childbearing potential not willing to use a double barrier method of contraception during the study and for 3 months following the last dose of study drug;
* Male patients whose sexual partner(s) are women of childbearing potential who are not willing to use a double barrier method of contraception, one of which includes a condom, during the study;
* Any of concurrent severe and/or uncontrolled medical condition, which could, in the opinion of the investigator, compromise participation in the study;
* Concurrent participation in another clinical study with an investigational medical product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Complete Molecular Response | At week 11 (acceptable window +2wks); after completion of two induction courses (1st Induction Course is 28 days) and before starting of the 1st Consolidation cycle at week 13
  Percentage of complete molecular responses after two cycles of induction therapy composed of a single cycle of blinatumomab followed by chemotherapy

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) response | End of blinatumomab infusion (End of the 1st Induction course which is 28 days); Day 40 of the study
  MRD response in bone marrow at the end of blinatumomab infusion (Induction cycle I)
Progression Free Survival (PFS) | Time from the day of CR/CRi documentation until the date of relapse, or death from any cause whichever came first, assessed up to 24 months
  Progression-free survival (PFS) in patients treated with blinatumomab followed by chemotherapy in the induction therapy
Overall Survival (OS) | Time between the start of leukemia-specific therapy (Day 1) until date of death of any cause, assessed up to 24 months
  Overall survival (OS) in patients treated with blinatumomab followed by chemotherapy in the induction therapy
AlloSCT | Week 18 ( after the completion of the 1st Consolidation cycle which is 21 days)
  Percentage of patients undergoing allogeneic stem cell transplantation (alloSCT) due to the suboptimal molecular response after blinatumomab and chemotherapy
Infectious complications during induction chemotherapy | At week 11; after completion of two induction courses (1st Induction Course is 28 days)
  Incidence of infectious complications during induction chemotherapy in patients treated with blinatumomab and chemotherapy
Incidence and severity of blinatumomab-related adverse events | At week 11; after completion of two induction courses (1st Induction Course is 28 days)
  incidence and severity of blinatumomab-related adverse events in the induction therapy

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Salek, MD, Principal Investigator — Institute of Hematology and Blood Transfusion, Czech Republic
Locations (5):
- Czechia (5):
  - University Hospital Brno, Internal hematology and oncology clinic, Brno
  - University Hospital Hradec Kralove,The 4th Department of Internal Medicine - Hematology, Hradec Králové
  - University Hospital Olomouc, Hematooncology Clinic, Olomouc
  - University Hospital Ostrava, Hematooncology Clinic, Ostrava
  - Institute of Hematology and Blood Transfusion, Czech Republic, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruggemann M, Schrauder A, Raff T, Pfeifer H, Dworzak M, Ottmann OG, Asnafi V, Baruchel A, Bassan R, Benoit Y, Biondi A, Cave H, Dombret H, Fielding AK, Foa R, Gokbuget N, Goldstone AH, Goulden N, Henze G, Hoelzer D, Janka-Schaub GE, Macintyre EA, Pieters R, Rambaldi A, Ribera JM, Schmiegelow K, Spinelli O, Stary J, von Stackelberg A, Kneba M, Schrappe M, van Dongen JJ; European Working Group for Adult Acute Lymphoblastic Leukemia (EWALL); International Berlin-Frankfurt-Munster Study Group (I-BFM-SG). Standardized MRD quantification in European ALL trials: proceedings of the Second International Symposium on MRD assessment in Kiel, Germany, 18-20 September 2008. Leukemia. 2010 Mar;24(3):521-35. doi: 10.1038/leu.2009.268. Epub 2009 Dec 24. PMID 20033054
- [Background] Kantarjian H, Stein A, Gokbuget N, Fielding AK, Schuh AC, Ribera JM, Wei A, Dombret H, Foa R, Bassan R, Arslan O, Sanz MA, Bergeron J, Demirkan F, Lech-Maranda E, Rambaldi A, Thomas X, Horst HA, Bruggemann M, Klapper W, Wood BL, Fleishman A, Nagorsen D, Holland C, Zimmerman Z, Topp MS. Blinatumomab versus Chemotherapy for Advanced Acute Lymphoblastic Leukemia. N Engl J Med. 2017 Mar 2;376(9):836-847. doi: 10.1056/NEJMoa1609783. PMID 28249141
- [Background] Mastrangelo R, Poplack D, Bleyer A, Riccardi R, Sather H, D'Angio G. Report and recommendations of the Rome workshop concerning poor-prognosis acute lymphoblastic leukemia in children: biologic bases for staging, stratification, and treatment. Med Pediatr Oncol. 1986;14(3):191-4. doi: 10.1002/mpo.2950140317. No abstract available. PMID 3528788
- [Background] Salek C, Folber F, Fronkova E, Prochazka B, Marinov I, Cetkovsky P, Mayer J, Doubek M; Czech Leukemia Study Group - for Life. Early MRD response as a prognostic factor in adult patients with acute lymphoblastic leukemia. Eur J Haematol. 2016 Mar;96(3):276-84. doi: 10.1111/ejh.12587. Epub 2015 Jun 22. PMID 25997106
- [Background] Topp MS, Gokbuget N, Stein AS, Zugmaier G, O'Brien S, Bargou RC, Dombret H, Fielding AK, Heffner L, Larson RA, Neumann S, Foa R, Litzow M, Ribera JM, Rambaldi A, Schiller G, Bruggemann M, Horst HA, Holland C, Jia C, Maniar T, Huber B, Nagorsen D, Forman SJ, Kantarjian HM. Safety and activity of blinatumomab for adult patients with relapsed or refractory B-precursor acute lymphoblastic leukaemia: a multicentre, single-arm, phase 2 study. Lancet Oncol. 2015 Jan;16(1):57-66. doi: 10.1016/S1470-2045(14)71170-2. Epub 2014 Dec 16. PMID 25524800
- [Background] Topp MS, Gokbuget N, Zugmaier G, Klappers P, Stelljes M, Neumann S, Viardot A, Marks R, Diedrich H, Faul C, Reichle A, Horst HA, Bruggemann M, Wessiepe D, Holland C, Alekar S, Mergen N, Einsele H, Hoelzer D, Bargou RC. Phase II trial of the anti-CD19 bispecific T cell-engager blinatumomab shows hematologic and molecular remissions in patients with relapsed or refractory B-precursor acute lymphoblastic leukemia. J Clin Oncol. 2014 Dec 20;32(36):4134-40. doi: 10.1200/JCO.2014.56.3247. Epub 2014 Nov 10. PMID 25385737
- [Background] Topp MS, Kufer P, Gokbuget N, Goebeler M, Klinger M, Neumann S, Horst HA, Raff T, Viardot A, Schmid M, Stelljes M, Schaich M, Degenhard E, Kohne-Volland R, Bruggemann M, Ottmann O, Pfeifer H, Burmeister T, Nagorsen D, Schmidt M, Lutterbuese R, Reinhardt C, Baeuerle PA, Kneba M, Einsele H, Riethmuller G, Hoelzer D, Zugmaier G, Bargou RC. Targeted therapy with the T-cell-engaging antibody blinatumomab of chemotherapy-refractory minimal residual disease in B-lineage acute lymphoblastic leukemia patients results in high response rate and prolonged leukemia-free survival. J Clin Oncol. 2011 Jun 20;29(18):2493-8. doi: 10.1200/JCO.2010.32.7270. Epub 2011 May 16. PMID 21576633
- [Background] van der Velden VH, Cazzaniga G, Schrauder A, Hancock J, Bader P, Panzer-Grumayer ER, Flohr T, Sutton R, Cave H, Madsen HO, Cayuela JM, Trka J, Eckert C, Foroni L, Zur Stadt U, Beldjord K, Raff T, van der Schoot CE, van Dongen JJ; European Study Group on MRD detection in ALL (ESG-MRD-ALL). Analysis of minimal residual disease by Ig/TCR gene rearrangements: guidelines for interpretation of real-time quantitative PCR data. Leukemia. 2007 Apr;21(4):604-11. doi: 10.1038/sj.leu.2404586. Epub 2007 Feb 8. PMID 17287850
- See also: Acute Lymphocytic Leukemia — https://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3aproject=medlineplus&v%3asources=...
- See also: Blinatumomab — https://druginfo.nlm.nih.gov/drugportal/name/blinatumomab